CLINICAL TRIAL: NCT04029961
Title: Pilot Study for the Development and Implementation of a Virtual Reality-based Radiation Therapy Education and Anxiety Mitigation Program
Brief Title: Virtual Reality Education Program to Reduce Anxiety During Radiation Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was suspended due to the COVID-19 pandemic. The study was then terminated to prevent inconsistencies in baseline anxiety for patients enrolled before vs after the COVID-19 pandemic.
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Marquette University (Other); Froedtert Hospital (Other)
Responsible Party: Principal Investigator, John LaDisa, Associate Professor, Biomedical Engineering, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PRO00032593
Record Dates: First submitted 2019-07-15; First posted 2019-07-23 (Actual); Results first posted 2021-05-10 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-04

CONDITIONS: Anxiety; Stress; Satisfaction, Patient; Preparedness; Information Needs
Keywords: Patient education; Virtual reality
MeSH Terms: conditions — Anxiety Disorders; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video Education (Active Comparator): Participants will receive video education on radiation therapy.
  Interventions: Other: Video Education
- VR-based Education (Experimental): Participants will receive VR-based education on radiation therapy.
  Interventions: Other: VR-based Education

INTERVENTIONS:
Other: Video Education — Prior to their CT simulation, participants will receive education on radiation therapy in the form of a video.
  Arms: Video Education
Other: VR-based Education — Prior to their CT simulation, participants will receive education on radiation therapy in the form of an immersive VR program delivered through a head-mounted display (HMD).
  Arms: VR-based Education

SUMMARY:
The purpose of this study is to compare the efficacy of an immersive virtual reality (VR)-based education program with a form of patient education commonly provided by clinics (e.g., an educational video) at delivering education to breast cancer patients as they prepare for radiation therapy treatment. Self-evaluation questionnaires completed by participants will be used to measure changes in information needs and anxiety, stress, preparedness and satisfaction levels pre/post education between the VR-based education and video education groups in this study. Expanded access to the current VR-based education program will depend on licensing status for associated assets by interested parties.

DETAILED DESCRIPTION:
Breast cancer patients experience anxiety, potentially reaching levels that are considered clinically-relevant. Prior research in this area has described the information needs of breast cancer patients at different time points as they proceed through the radiotherapy treatment process. Of high importance seems to be addressing patients' information needs through sensory and procedural information as a mechanism of anxiety reduction.

The study team created an immersive VR-based education program that enables breast cancer patients to experience the procedure and emotions associated with radiation therapy prior to their actual treatment by offering controlled virtual exposure to the clinical environments involved in the treatment process. An educational video on the process of receiving radiation therapy is considered standard education at the majority of the clinical sites involved in this study.

Participants enrolled in this study will be randomly assigned to either the VR-based education group or the video education group. Participation in this project will provide insight into aspects of patient education that are most effective at reducing anxiety and stress levels and meeting patients' information needs when undergoing radiation therapy treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is 18 years of age or older
2. Patient is female
3. Patient has been diagnosed with breast cancer
4. Patient will be receiving whole breast radiation therapy without supraclavicular nodal irradiation
5. Patient is scheduled for an outpatient radiation oncology visit
6. Patient has the ability to understand a written informed consent document, and the willingness to sign it
7. Patient has the ability to complete a series of self-reported questionnaires

Exclusion Criteria:

1. Non-English-speaking patients (as the VR education program includes English narration)
2. Patients with visual defects that affect their ability to watch a movie
3. Patients with auditory defects that affect their ability to listen with headphones
4. Patients who have worked in the field of radiation oncology as they would have previously undergone treatment-related education
5. Patients who have been treated previously with radiation oncology as they would have previously undergone treatment-related education
6. Patients that have been diagnosed with epilepsy, conditions causing seizures, or have any previous history of seizures because a very minute number of head-mounted display (HMD) users have experienced a seizure as a result of using the device
7. Patients with a reported history of cognitive disability as their ability to understand educational content may be impaired
8. Patients with a history of severe motion sickness because a side effect of using a HMD in a very small number of users is motion sickness symptoms
9. Patients with a pacemaker, hearing aid(s), and/or defibrillator, while patients with other types of electronic medical devices / implants will be assessed for eligibility on a case-by-case basis because there could be potential interference with the HMD

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2020-04-14 (Actual); Study Completion 2020-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John LaDisa, PhD, Principal Investigator — Medical College of Wisconsin; Monica Shukla, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert & the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Halkett GK, Kristjanson LJ, Lobb E, Little J, Shaw T, Taylor M, Spry N. Information needs and preferences of women as they proceed through radiotherapy for breast cancer. Patient Educ Couns. 2012 Mar;86(3):396-404. doi: 10.1016/j.pec.2011.05.010. Epub 2011 Jun 12. PMID 21664788
- [Background] Bekelis K, Calnan D, Simmons N, MacKenzie TA, Kakoulides G. Effect of an Immersive Preoperative Virtual Reality Experience on Patient Reported Outcomes: A Randomized Controlled Trial. Ann Surg. 2017 Jun;265(6):1068-1073. doi: 10.1097/SLA.0000000000002094. PMID 27906757
- [Background] Halkett GK, Kristjanson LJ. Validity and reliability testing of two instruments to measure breast cancer patients' concerns and information needs relating to radiation therapy. Radiat Oncol. 2007 Nov 25;2:43. doi: 10.1186/1748-717X-2-43. PMID 18036247
- [Background] Spielberger, C. State-Trait Anxiety Inventory for Adults - Manual, Instrument and Scoring Guide. 2015 Consulting Psychologists Press, Inc. Mind Garden, Inc.
- See also: Patient Video by the American Society for Therapeutic Radiation Oncology (ASTRO) — https://www.rtanswers.org/What-is-Radiation-Therapy/What-to-Expect

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on screening pre-existing medical records conducted by the study team/staff and physician concurrence at 3 academic medical centers within the same regional health network between July 2019 and March 2020. The first participant was enrolled in August 2019 and the last participant was enrolled in March 2020.
Pre-assignment Details: Of 28 consented participants, 26 were found eligible and randomized to an intervention. One participant was considered ineligible after consent after moving treatment out of state and one participant's participation in the study was cancelled due to the COVID-19 pandemic.
Period: Overall Study
Arm/Group | Video Education | VR-based Education
Started | 13 | 13
Completed | 12 | 12
Not Completed | 1 | 1
Not completed — Withdrawal after participant advisal they viewed exact same education intervention prior to visit | 1 | 0
Not completed — Change in Treatment Course | 0 | 1

BASELINE CHARACTERISTICS:
Population: Only complete datasets were analyzed in this study. There was one participant in the VR arm for whom baseline measurements were collected, but not used in the final data analysis, as the patient was withdrawn due to a change in treatment course prior to completing the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Video Education | VR-based Education | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.25 (9.00) | 58.92 (9.29) | 58.08 (8.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Non-Hispanic | 12 | 12 | 24
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 12 | 24
Previous chemotherapy = yes [Count of Participants; unit: Participants] | 3 | 2 | 5
T stage = non-DCIS [Count of Participants; unit: Participants] — The T stage within the TNM Cancer staging system provides information on the tumor. DCIS is ductal carcinoma in situ, a non-invasive or pre-invasive cancer.
  Participants | 9 | 10 | 19
Highest education level = high school/GED [Count of Participants; unit: Participants] | 3 | 3 | 6
Study site = Group 1 [Count of Participants; unit: Participants] — Study sites were grouped based on similarity in clinical workflow, to be incorporated as a covariate in the statistical models. Patient numbers enrolled at each specific study site or within specific groups are purposefully not provided for patient confidentiality purposes, hence the generic naming convention of "group 1" instead of clinic name(s).
  Participants | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Intra- and Inter-arm Differences in Pre-post Intervention Changes in Anxiety Using the State Trait Anxiety Inventory (STAI) for Adults Scores
Description: The STAI was administered as a self-evaluation questionnaire at three time points. The STAI consists of two scales: one for measuring trait anxiety and one for measuring state anxiety. Both of the scales have ranges from 20 - 80, with higher scores representing higher anxiety.
Time Frame: Directly pre/post education (education appointment), directly following first radiation therapy (RT) treatment (first RT session)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Video Education | VR-based Education
Number analyzed (Participants) | 12 | 12
score on a scale
  STAI-Trait: Pre-education | 34.17 (9.504) | 32.75 (5.083)
  STAI-State: Pre-education | 35.42 (8.118) | 37.17 (8.943)
  STAI-State: Post-education | 29.58 (9.434) | 31.92 (6.908)
  STAI-State: After radiation therapy | 33.00 (10.41) | 31.00 (7.897)
Statistical Analysis 1: Comparison: Video Education vs VR-based Education; Test type: Other — Multivariate regression model and intra-arm differences in measure scores between time points; p < 0.05, multivariate regression — Multivariate regression was adjusted for covariates of study site, highest education level, prior chemotherapy, age, & T stage. Random effects was adjusted for multiple measurements. Multiplicity corrections were conducted via Holm-Sidak method

2. Primary Outcome: Intra- and Inter-arm Differences in Pre-post Intervention Changes in Stress Using the Visual Analog Scale for Stress Scores
Description: The Visual Analog Scale for Stress was administered as a self-evaluation questionnaire at three time points. Participants indicated where they fell in terms of stress level from 0 (no stress at all) to 100 (most stressed ever).
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Video Education | VR-based Education
Number analyzed (Participants) | 12 | 12
score on a scale
  Pre-education | 25.17 (19.85) | 35.83 (21.41)
  Post-education | 22.83 (22.93) | 22.50 (17.25)
  After radiation therapy | 33.08 (30.70) | 25.83 (18.69)
Statistical Analysis 1: Comparison: Video Education vs VR-based Education; Test type: Other — Multivariate regression model and intra-arm differences in measure scores between time points; p < 0.05, multivariate regression — [p-value comment as in outcome 1, analysis 1]

3. Primary Outcome: Intra- and Inter-arm Differences in Pre-post Intervention Changes in Preparedness Using the Visual Analog Scale for Preparedness Scores
Description: The Visual Analog Scale for Preparedness was administered as a self-evaluation questionnaire at three time points. Participants indicated where they fell in terms of preparedness for their RT treatment from 0 (not prepared at all) to 100 (completely prepared).
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Video Education | VR-based Education
Number analyzed (Participants) | 12 | 12
score on a scale
  Pre-education | 63.50 (22.11) | 51.25 (22.37)
  Post-education | 82.50 (21.73) | 82.42 (14.59)
  After radiation therapy | 90.83 (11.04) | 87.08 (19.36)
Statistical Analysis 1: Comparison: Video Education vs VR-based Education; Test type: Other — Multivariate regression model and intra-arm differences in measure scores between time points; p < 0.05, multivariate regression — [p-value comment as in outcome 1, analysis 1]

4. Primary Outcome: Intra- and Inter-arm Differences in Pre-post Intervention Changes in Satisfaction Using the Visual Analog Scale for Satisfaction Scores
Description: The Visual Analog Scale for Satisfaction was administered at three time points. Participants indicated where they fell in terms of satisfaction from their experience with the radiation oncology department from 0 (not satisfied at all) to 100 (completely satisfied).
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Video Education | VR-based Education
Number analyzed (Participants) | 12 | 12
score on a scale
  Pre-education | 95.42 (6.557) | 87.92 (11.96)
  Post-education | 95.42 (6.557) | 91.25 (10.03)
  After radiation therapy | 95.83 (9.003) | 89.17 (19.64)
Statistical Analysis 1: Comparison: Video Education vs VR-based Education; Test type: Other — Multivariate regression model and intra-arm differences in measure scores between time points; p < 0.05, multivariate regression — [p-value comment as in outcome 1, analysis 1]

5. Primary Outcome: Proportional Differences in Pre-post Intervention Changes in the "Met" Need Count Per Arm of Information Need Topics Related to Radiation Therapy Treatment Using the Information Needs Scale Scores
Description: The Information Needs Scale was administered as a self-evaluation questionnaire at three time points. Participants were asked to indicate how important it was for them to have information on a set of items related to radiation therapy treatment from 1 (not important) to 9 (very important). Participants were also asked to indicate whether they felt their needed level of information for each item was met, partially met, or unmet at the time of questionnaire completion, which is reported here.
Time Frame: as for outcome 1
Population: Proportional differences in pre-post intervention changes in the "met" need count per arm of information need topics related to radiation therapy treatment using the Information Needs Scale scores.
Measure: Count of Participants; unit: Participants
Arm/Group | Video Education | VR-based Education
Number analyzed (Participants) | 12 | 12
Participants
  Pre-education: 1. Why I need to receive radiation therapy | 6 | 9
  Pre-education: 2. What radiation therapy will involve | 5 | 1
  Pre-education: 3. What happens during the planning appointment | 3 | 1
  Pre-education: 4. How my treatment is planned | 5 | 1
  Pre-education: 5. The radiation oncologist who will be treating me | 11 | 8
  Pre-education: 6. The roles of the different staff in the department | 4 | 2
  Pre-education: 7. How much of my breast will be treated | 3 | 2
  Pre-education: 8. The treatment machine | 1 | 1
  Pre-education: 9. What happens on the first day | 0 | 1
  Pre-education: 10. Why there are cameras & computers in treatment room & what are they for | 0 | 2
  Pre-education: 11. What the x-rays that are taken on the treatment machine are used for | 1 | 0
  Pre-education: 12. What side effects I may experience | 3 | 1
  Pre-education: 13. Whether the radiation will effect my heart | 7 | 0
  Pre-education: 14. Whether my lungs will be damaged by treatment | 6 | 0
  Pre-education: 15. Other people's experiences of receiving treatment | 3 | 0
  Pre-education: 16. How to take care of my skin | 2 | 1
  Pre-education: 17. Whether I can keep working during treatment | 3 | 3
  Pre-education: 18. Who can provide me with information | 7 | 2
  Pre-education: 19. What will happen after treatment is finished | 1 | 0
  Pre-education: 20. The cost of treatment | 3 | 0
  Pre-education: 21. Transport that is available | 3 | 0
  Pre-education: 22. Parking | 7 | 3
  Post-education: 1. Why I need to receive radiation therapy | 10 | 11
  Post-education: 2. What radiation therapy will involve | 10 | 11
  Post-education: 3. What happens during the planning appointment | 10 | 11
  Post-education: 4. How my treatment is planned | 11 | 10
  Post-education: 5. The radiation oncologist who will be treating me | 12 | 9
  Post-education: 6. The roles of the different staff in the department | 11 | 10
  Post-education: 7. How much of my breast will be treated | 5 | 6
  Post-education: 8. The treatment machine | 11 | 11
  Post-education: 9. What happens on the first day | 11 | 10
  Post-education: 10. Why there are cameras & computers in treatment room & what are they for | 11 | 9
  Post-education: 11. What the x-rays that are taken on the treatment machine are used for | 11 | 10
  Post-education: 12. What side effects I may experience | 8 | 10
  Post-education: 13. Whether the radiation will effect my heart | 8 | 7
  Post-education: 14. Whether my lungs will be damaged by treatment | 8 | 7
  Post-education: 15. Other people's experiences of receiving treatment | 11 | 4
  Post-education: 16. How to take care of my skin | 6 | 2
  Post-education: 17. Whether I can keep working during treatment | 9 | 10
  Post-education: 18. Who can provide me with information | 11 | 10
  Post-education: 19. What will happen after treatment is finished | 10 | 4
  Post-education: 20. The cost of treatment | 2 | 1
  Post-education: 21. Transport that is available | 6 | 0
  Post-education: 22. Parking | 8 | 1
  After radiation therapy: 1. Why I need to receive radiation therapy | 10 | 12
  After radiation therapy: 2. What radiation therapy will involve | 10 | 12
  After radiation therapy: 3. What happens during the planning appointment | 11 | 12
  After radiation therapy: 4. How my treatment is planned | 11 | 11
  After radiation therapy: 5. The radiation oncologist who will be treating me | 12 | 12
  After radiation therapy: 6. The roles of the different staff in the department | 11 | 12
  After radiation therapy: 7. How much of my breast will be treated | 10 | 11
  After radiation therapy: 8. The treatment machine | 11 | 12
  After radiation therapy: 9. What happens on the first day | 11 | 11
  After radiation therapy: 10. Why there are cameras & computers in treatment room & what are they for | 10 | 12
  After radiation therapy: 11. What the x-rays that are taken on the treatment machine are used for | 9 | 9
  After radiation therapy: 12. What side effects I may experience | 9 | 8
  After radiation therapy: 13. Whether the radiation will effect my heart | 8 | 10
  After radiation therapy: 14. Whether my lungs will be damaged by treatment | 9 | 10
  After radiation therapy: 15. Other people's experiences of receiving treatment | 8 | 7
  After radiation therapy: 16. How to take care of my skin | 5 | 6
  After radiation therapy: 17. Whether I can keep working during treatment | 8 | 9
  After radiation therapy: 18. Who can provide me with information | 12 | 11
  After radiation therapy: 19. What will happen after treatment is finished | 9 | 6
  After radiation therapy: 20. The cost of treatment | 5 | 3
  After radiation therapy: 21. Transport that is available | 6 | 3
  After radiation therapy: 22. Parking | 6 | 3
Statistical Analysis 1: Comparison: Video Education vs VR-based Education; The statistical test described below was only performed on the top 10 items on the scale rated the highest in importance by participants. The top 10 items were determined by computing the mean rating for each item (participants gave each item a rating from '1' - '9' with higher values representing greater importance) and selecting the 10 items with the largest mean values, excluding the item "the radiation oncologist who will be treating me" as that item was not addressed in either intervention; Test type: Other — A univariate analysis comparing the proportion of each arm that indicated an item was "met," evaluated for each item at each time point; p < 0.05, Univariate analysis

ADVERSE EVENTS:
Time Frame: 32 weeks
Arm/Group | Video Education | VR-based Education
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

LIMITATIONS AND CAVEATS:
This study is based on aggregate data from a small sample size. There were elements of this study difficult to standardize, such as educational information patients acquired on RT from other sources.

The Information Needs Scale instructions could be interpreted two ways. It became unclear later on in the study whether patients should have been rating items based on overall informational importance or current need to obtain information. Patients may have completed this portion differently.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-06-14): https://cdn.clinicaltrials.gov/large-docs/61/NCT04029961/Prot_SAP_000.pdf
  • Informed Consent Form (2019-06-15): https://cdn.clinicaltrials.gov/large-docs/61/NCT04029961/ICF_001.pdf